CLINICAL TRIAL: NCT00960297
Title: Phase II Trial of Preoperative Chemotherapy and Bevacizumab in Patients With Stage IB (>4 cm), II, or Select Stage III Non-Small Cell Lung Cancer
Brief Title: Preoperative Chemotherapy and Bevacizumab in Patients With Stage IB (>4 cm), II, or Select Stage III NSCLC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to slow accrual
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LUN 144
Record Dates: First submitted 2009-08-13; First posted 2009-08-17 (Estimated); Results first posted 2013-11-08 (Estimated); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; NSCLC; Preoperative chemotherapy; Bevacizumab; Avastin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Carboplatin/Paclitaxel/Bevacizumab (Experimental): Preoperative chemotherapy and bevacizumab
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Bevacizumab

INTERVENTIONS:
Drug: Carboplatin — Carboplatin: AUC=6, given IV on Days 1, 22, 43, and 64
  Other Names: Paraplatin
Drug: Paclitaxel — Paclitaxel: 200 mg/m2, given IV on Days 1, 22, 43, and 64
  Other Names: Taxol
Drug: Bevacizumab — Bevacizumab: 15 mg/kg, given IV on Days 1, 22, and 43 (Note: bevacizumab will not be dosed on Day 64 prior to surgery)
  Other Names: Avastin

SUMMARY:
The rationale for this multicenter, phase II trial is to examine the impact of carboplatin/paclitaxel with bevacizumab in the preoperative treatment of patients with stage IB (> 4.0 cm), II, and select stage III NSCLC. If this novel regimen proves to be safe and active in this setting, this would provide rationale for further investigation in a larger, prospective, randomized setting.

DETAILED DESCRIPTION:
Adjuvant chemotherapy for patients with completely resected stage II and select stage III NSCLC is considered standard therapy. At least three large, prospective randomized trials have proven the benefit of adjuvant chemotherapy in improving survival in these patients (with a magnitude of benefit ranging from 4-12%). However, in patients who are not considered to be candidates for up-front complete resection, preoperative therapy may be indicated. Many of these patients will subsequently be eligible for resection (bimodality therapy). The rationale for this multicenter, Phase II trial is to examine the impact of carboplatin/paclitaxel with bevacizumab in the preoperative treatment of patients with stage IB (>4.0 cm), II, and select stage III NSCLC. This trial will be conducted by the Sarah Cannon Research Institute Oncology Research Consortium. If this novel regimen proves to be safe and active in this setting, this would provide rationale for further investigation in a larger, prospective, randomized setting.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18 years.
2. Histologically-confirmed NSCLC (adenocarcinoma, large cell, and undifferentiated). Patients with squamous histology are not eligible.
3. Life expectancy of at least 12 weeks.
4. Patients with the following stages of NSCLC:

   * T2 N0 tumors: Limited to tumors >=4 cm.
   * T1-2 N1 tumors.
   * T3 N0-1 tumors (excluding superior sulcus tumors): Including tumors involving the chest wall, proximal airway, or mediastinal pleura where preoperative RT is not planned.
   * T1-2 N2 tumors: For patients with N2 disease involving 1 zone (Upper zone (R), AP zone (L), subcarinal zone, or lower zone) and nodes <=2 cm in diameter.
   * T4 N0-1 tumors (excluding superior sulcus tumors): T4 lesions, other than malignant effusions where radiotherapy is not planned.
5. Patients with clinical N2 involvement must have histologic confirmation by mediastinoscopy (or alternate biopsy procedure).
6. Tumors should be considered potentially resectable.
7. No evidence of extrathoracic metastatic disease.
8. Patients must have measurable disease by RECIST version 1.1 criteria.
9. Patients must be candidates (medically) for chemotherapy followed by surgical resection.
10. Adequate recovery from recent surgery. At least 1 week must have elapsed from the time of a minor surgery (with the exception of portacath or other central access catheter placement); at least 4 weeks must have elapsed from the time of a major surgery.
11. Laboratory values as follows:

    * Absolute neutrophil count (ANC) >=1500/µL
    * Hemoglobin (Hgb) >=9 g/dL
    * Platelets >=100,000/uL
    * AST/SGOT and ALT/SGPT within normal limits (WNL)
    * Total bilirubin within normal limits (WNL)
    * Creatinine <=1.5 mg/dL
12. ECOG Performance Status grade 0 or 1.
13. Women of childbearing potential must have a negative serum or urine pregnancy test performed within 7 days prior to start of treatment. Women of childbearing potential or men with partners of childbearing potential must use effective birth control measures during treatment. If a woman becomes pregnant or suspects she is pregnant while participating in this study, she must agree to inform her treating physician immediately.
14. Patient must be accessible for treatment and follow-up.
15. Patients must be able to understand the investigational nature of this study and give written informed consent prior to study entry.

Exclusion Criteria:

1. Mixed small-cell and non-small cell histologies.
2. Pulmonary carcinoid tumors.
3. History of prior malignancy within 3 years, with the exception of non-melanoma skin cancer or carcinoma in situ.
4. Peripheral neuropathy >= grade 1.
5. Patients receiving thrombolytic therapy within 10 days of starting study treatment are ineligible. Therapeutic anticoagulation is allowed if the anticoagulant dosing is stable.
6. History of acute myocardial infarction or unstable angina within 6 months prior to Day 1 of study treatment.
7. History of or stroke or ischemic attack within 6 months prior to Day 1 of study treatment.
8. Inadequately controlled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg) in spite of medical management.
9. New York Heart Association (NYHA) class II or greater congestive heart failure (CHF).
10. Patients with significant vascular disease (e.g., aortic aneurysm requiring surgical repair, or recent peripheral arterial thrombosis) within 6 months prior to Day 1 of study treatment.
11. Any prior history of hypertensive crisis or hypertensive encephalopathy.
12. Patients with hematemesis or hemoptysis (>=1/2 teaspoon of bright red blood per episode) within 1 month prior to Day 1 of study treatment.
13. Proteinuria at screening, as demonstrated by either:

    * Urine protein: creatinine (UPC) ratio >=1.0 (see Appendix A) at screening, or
    * Urine dipstick for proteinuria >=2+ (patients discovered to have >=2+ proteinuria on dipstick analysis should undergo a 24-hour urine collection and must have <=1g of protein in 24 hours to be eligible).
14. Patients with a serious non-healing wound, active ulcer, or untreated bone fracture.
15. Patients with evidence of bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation).
16. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 1 of study treatment.
17. Women who are pregnant (positive pregnancy test) or lactating.
18. Use of any non-approved or investigational agent within 28 days of administration of the first dose of study drug.
19. Patients may not receive any other investigational or anti-cancer treatments while participating in this study.
20. Concurrent severe, intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.
21. History of hypersensitivity to active or inactive excipients of any component of treatment.
22. Inability to comply with study and/or follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-08; Primary Completion 2012-11 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Spigel, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (6):
- United States (6):
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Providence Medical Group, Terre Haute, Indiana
  - Norton Cancer Institute, Louisville, Kentucky
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Tennessee Oncology, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- Carboplatin/Paclitaxel/Bevacizumab: Preoperative chemotherapy and bevacizumab
  Bevacizumab : Bevacizumab: 15 mg/kg, given IV on Days 1, 22, and 43 (Note: bevacizumab will not be dosed on Day 64 prior to surgery)
  Paclitaxel : Paclitaxel: 200 mg/m2, given IV on Days 1, 22, 43, and 64
  Carboplatin : Carboplatin: AUC=6, given IV on Days 1, 22, 43, and 64
Period: Overall Study
Arm/Group | Carboplatin/Paclitaxel/Bevacizumab
Started | 4
Completed | 1
Not Completed | 3
Not completed — Physician Decision | 1
Not completed — Venous port infection | 1
Not completed — Disease progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | Carboplatin/Paclitaxel/Bevacizumab
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: To Assess 3-year Overall Survival in Patients With Stage IB (>4.0 cm), II, or Select Stage III NSCLC Treated With Preoperative Carboplatin, Paclitaxel, and Bevacizumab Followed by Surgical Resection.
Time Frame: 36 months
Population: Study ended early due to slow accrual.
Arm/Group | Carboplatin/Paclitaxel/Bevacizumab
Number analyzed (Participants) | 0

2. Secondary Outcome: Clinical & Pathologic Response Rate
Time Frame: 60 months
Population: Results were not analyzed as the study ended early due to slow accrual and incomplete data collection
Arm/Group | Carboplatin/Paclitaxel/Bevacizumab
Number analyzed (Participants) | 0

3. Secondary Outcome: Complete Resection Rate
Time Frame: 60 months
Population: Results were not analyzed as the study ended early due to slow accrual and incomplete data collection.
Arm/Group | Carboplatin/Paclitaxel/Bevacizumab
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants Experiencing Adverse Events as a Measure of Toxicity
Description: An adverse event (AE) is the development of an undesirable medical condition, or the deterioration of a preexisting medical condition (other than the condition that is being treated by the trial) following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. The number of participants experiencing such adverse events are reported here.
Time Frame: 45 months
Measure: Count of Participants; unit: Participants
Arm/Group | Carboplatin/Paclitaxel/Bevacizumab
Number analyzed (Participants) | 4
Participants | 4

5. Secondary Outcome: Progression-free Survival
Time Frame: 60 months
Population: Results were not analyzed as the study ended early due to slow accrual and incomplete data collection.
Arm/Group | Carboplatin/Paclitaxel/Bevacizumab
Number analyzed (Participants) | 0

6. Secondary Outcome: Overall Survival
Time Frame: 60 months
Population: Results were not analyzed as the study ended early due to slow accrual and incomplete data collection.
Arm/Group | Carboplatin/Paclitaxel/Bevacizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Carboplatin/Paclitaxel/Bevacizumab
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin/Paclitaxel/Bevacizumab (N=4)
Colitis, nonspecific (Gastrointestinal disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin/Paclitaxel/Bevacizumab (N=4)
Abdominal distension - mild (Gastrointestinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
alkaline phosporus (L) (Metabolism and nutrition disorders) | 1 (1)
Altered mental status (Nervous system disorders) | 1 (1)
ANC (Blood and lymphatic system disorders) | 1 (3)
Anorexia (Endocrine disorders) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Chapped lips (Skin and subcutaneous tissue disorders) | 1 (1)
Chloride, low (Metabolism and nutrition disorders) | 2 (2)
CO2 (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Coarse crackles, right lung base (Respiratory, thoracic and mediastinal disorders) | 1 (1)
cold sensitivity (General disorders) | 1 (1)
Colitis, nonspecific (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Creatinine (Metabolism and nutrition disorders) | 2 (3)
Dark Stools (Gastrointestinal disorders) | 1 (1)
Dehisce, port site (Skin and subcutaneous tissue disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Diminished breath sounds (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Dizziness (Nervous system disorders) | 1 (1)
Edema (General disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Failute to thrive (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Febrile neutropenia (Infections and infestations) | 1 (1)
Fever (Infections and infestations) | 2 (3)
Gaseous (Gastrointestinal disorders) | 1 (1)
Body Aches, generalized (General disorders) | 1 (1)
HCT, low (Blood and lymphatic system disorders) | 1 (1)
Head Cold (Respiratory, thoracic and mediastinal disorders) | 1 (1)
headache (General disorders) | 1 (1)
Hematologic, ANC (Blood and lymphatic system disorders) | 2 (3)
Hematologic, Hemoglobin (Blood and lymphatic system disorders) | 4 (9)
Hematologic, platelets (Blood and lymphatic system disorders) | 2 (5)
Hematologic, WBC (Blood and lymphatic system disorders) | 3 (7)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 2 (4)
hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
hypertension (Vascular disorders) | 1 (1)
hypoalbuminemia (Metabolism and nutrition disorders) | 2 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (3)
hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
infection (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 2 (2)
Malaise (General disorders) | 1 (1)
Mental Status Change (Psychiatric disorders) | 1 (1)
Mucositis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (3)
Neuropathy (Nervous system disorders) | 2 (2)
Orthostasis (Vascular disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 1 (8)
Proteinuria (Renal and urinary disorders) | 2 (4)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal insufficiency (Renal and urinary disorders) | 1 (1)
Rigors (General disorders) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Soreness, port site (General disorders) | 1 (1)
Purulent Drainage (General disorders) | 1 (1)
thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Bilirubin (Investigations) | 2 (2)
Total Protein (Renal and urinary disorders) | 1 (4)
Urine Protein Creatinine Ratio (Renal and urinary disorders) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Weakness (Musculoskeletal and connective tissue disorders) | 4 (4)
Weightloss (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.